CLINICAL TRIAL: NCT00114179
Title: A Phase II Study of Bevacizumab With Concurrent Capecitabine and Radiation Followed by Maintenance Gemcitabine and Bevacizumab For Locally Advanced Pancreatic Cancer
Brief Title: Capecitabine, Bevacizumab, and Radiation Therapy Followed By Gemcitabine and Bevacizumab in Treating Patients With Locally Advanced Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02661; NCI-2012-02661 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000434846; RTOG-0411 (Other: Radiation Therapy Oncology Group); RTOG-0411 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Adenocarcinoma of the Pancreas; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Radiotherapy; Radiation; Bevacizumab; Gemcitabine

ARMS (1):
- Treatment (capecitabine, radiation, bevacizumab, gemcitabine) (Experimental): Chemoradiotherapy and bevacizumab: Patients receive oral capecitabine twice daily and undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38. Patients also receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29. Patients undergo reevaluation 3-4 weeks after completion of chemoradiotherapy and bevacizumab.
  Patients with no evidence of disease progression proceed to maintenance therapy. Patients with a marked response may undergo surgery at the discretion of the attending surgeon and then proceed to maintenance therapy approximately 4-8 weeks later.
  Maintenance therapy: Beginning within 4-7 weeks after completion of chemoradiotherapy and bevacizumab, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30 minutes on days 1 and 15 provided that blood counts have returned to normal. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Radiation: radiation therapy; Biological: bevacizumab; Procedure: therapeutic conventional surgery; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Procedure: therapeutic conventional surgery — Undergo surgery
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar

SUMMARY:
Drugs used in chemotherapy, such as capecitabine and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Capecitabine may make tumor cells more sensitive to radiation therapy. Bevacizumab may make tumor cells more sensitive to both chemotherapy and radiation therapy. Giving chemotherapy and bevacizumab before and after radiation therapy may kill more tumor cells. This phase II trial is studying how well giving capecitabine and bevacizumab together with radiation therapy followed by gemcitabine and bevacizumab works in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare 1-year overall survival of patients with unresectable locally advanced pancreatic cancer treated with capecitabine, bevacizumab, and radiotherapy followed by maintenance therapy comprising gemcitabine and bevacizumab to a historical control.

SECONDARY OBJECTIVES:

I. Determine the frequency of serious unacceptable adverse events in patients treated with this regimen.

II. Determine the response rate in patients treated with this regimen. III. Determine the progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Chemoradiotherapy and bevacizumab: Patients receive oral capecitabine twice daily and undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38. Patients also receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29. Patients undergo reevaluation 3-4 weeks after completion of chemoradiotherapy and bevacizumab.

Patients with no evidence of disease progression proceed to maintenance therapy. Patients with a marked response may undergo surgery at the discretion of the attending surgeon and then proceed to maintenance therapy approximately 4-8 weeks later.

Maintenance therapy: Beginning within 4-7 weeks after completion of chemoradiotherapy and bevacizumab, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30 minutes on days 1 and 15 provided that blood counts have returned to normal. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for survival.

PROJECTED ACCRUAL: A total of 82 patients will be accrued for this study within 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas

  * Locally advanced disease
  * Unresectable disease
* All malignant disease must be encompassable within a single irradiation field
* Radiographically assessable disease
* Patients with biliary or gastroduodenal obstruction are eligible provided drainage or surgical bypass was performed prior to initiation of study treatment
* No evidence of gastric outlet obstruction
* No evidence of duodenal invasion on CT scan
* No evidence of metastatic disease in the major viscera
* No peritoneal seeding or ascites
* Performance status - Zubrod 0-1
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No evidence of bleeding diathesis
* ALT < 3 times upper limit of normal
* Bilirubin < 2.0 mg/dL
* INR ≤ 1.5
* No evidence of coagulopathy
* Creatinine clearance > 50 mL/min
* Urine protein < 1,000 mg by 24-hour urine collection (for patients with proteinuria ≥ 1+ by dipstick or urinalysis OR urine protein:creatinine ratio ≥ 1.0)
* No myocardial infarction within the past 6 months
* No unstable angina within the past 6 months
* No arterial thromboembolic events within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Clinically significant peripheral artery disease
* No unstable symptomatic arrhythmia requiring medication (e.g., chronic atrial arrhythmia [i.e., atrial fibrillation or paroxysmal supraventricular tachycardia])

  * Patients with an atrial arrhythmia are eligible provided the condition is well controlled on stable medication
* No New York Heart Association class II-IV congestive heart failure
* No history of arteriovenous malformation
* No history of aneurysm
* No uncontrolled hypertension (i.e., blood pressure > 160/90 mm Hg with medication)
* No other clinically significant cardiac disease
* No AIDS
* No significant infection
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Not pregnant
* No nursing during and for ≥ 3-4 months after completion of study treatment
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3-4 months after completion of study treatment
* No history of gastrointestinal fistula or perforation
* No other malignancy within the past two years except nonmelanoma skin cancer or carcinoma in situ of the cervix, uterus, or bladder
* No significant traumatic injury within the past 4 weeks
* No serious nonhealing wound or ulcer
* No current healing fracture
* No known or suspected dihydropyrimidine dehydrogenase deficiency
* No other medical condition that would preclude study participation
* No concurrent interleukin-11
* No prior chemotherapy for pancreatic cancer
* More than 2 years since prior chemotherapy for another malignancy
* No prior radiotherapy to the planned irradiation field
* No concurrent intensity modulated radiotherapy
* No other concurrent radiotherapy
* See Disease Characteristics
* More than 4 weeks since prior major surgical procedure or open biopsy
* More than 1 week since prior fine needle aspiration or core biopsy
* No prior organ transplantation
* No concurrent major surgical procedure
* More than 30 days since prior and no concurrent cimetidine

  * Concurrent ranitidine or a drug from another anti-ulcer class allowed
* More than 4 weeks since prior and no concurrent sorivudine or brivudine
* No concurrent warfarin during chemoradiotherapy

  * Concurrent warfarin allowed beginning 2 weeks after completion of chemoradiotherapy
  * Concurrent low molecular weight heparin allowed (at any time during study participation)
* No other concurrent investigational agents
* No other concurrent cytotoxic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 1 year
  Will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Frequency of patients developing grade 3 or greater adverse events as defined per CTCAE version 3.0 | Up to 1 year
Progression-free survival | Up to 1 year
  Will be estimated using the Kaplan-Meier method.
Response rate | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Crane, Principal Investigator — Radiation Therapy Oncology Group
Locations (1):
- Radiation Therapy Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Crane CH, Winter K, Regine WF, Safran H, Rich TA, Curran W, Wolff RA, Willett CG. Phase II study of bevacizumab with concurrent capecitabine and radiation followed by maintenance gemcitabine and bevacizumab for locally advanced pancreatic cancer: Radiation Therapy Oncology Group RTOG 0411. J Clin Oncol. 2009 Sep 1;27(25):4096-102. doi: 10.1200/JCO.2009.21.8529. Epub 2009 Jul 27. PMID 19636002